CLINICAL TRIAL: NCT04372186
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Tocilizumab in Hospitalized Patients With COVID-19 Pneumonia
Brief Title: A Study to Evaluate the Efficacy and Safety of Tocilizumab in Hospitalized Participants With COVID-19 Pneumonia
Acronym: EMPACTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML42528
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Results first posted 2021-09-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive one intravenous (IV) infusion of placebo, in addition to SOC. Up to one additional infusion may be given.
  Interventions: Drug: Placebo
- Tocilizumab (Experimental): Participants will receive one IV infusion of TCZ in addition to SOC. Up to one additional infusion may be given.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Placebo — Participants will receive one dose of IV placebo matched to TCZ. Up to one additional dose may be given.
  Arms: Placebo
Drug: Tocilizumab — Participants will receive one IV infusion of TCZ 8 mg/kg, with a maximum dose of 800 mg. Up to one additional dose may be given.
  Arms: Tocilizumab

SUMMARY:
This study (EMPACTA) will a) evaluate the efficacy and safety of tocilizumab (TCZ) compared with a placebo in combination with standard of care (SOC) in hospitalized participants with COVID-19 pneumonia, and b) include an optional long-term extension for eligible participants to explore the long-term sequelae of resolved COVID-19 pneumonia.

ELIGIBILITY:
Inclusion Criteria

* Hospitalized
* COVID-19 pneumonia confirmed by a positive polymerase chain reaction (PCR) of any specimen and radiographic imaging
* SpO2 < 94% while on ambient air

Inclusion Criteria Specific to Long-Term Extension

* Participated in Study ML42528 (EMPACTA) (includes participants who completed or discontinued early from the main study)

Exclusion Criteria

* Known severe allergic reactions to TCZ or other monoclonal antibodies
* Require continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP), or invasive mechanical ventilation
* Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments
* Immunocompromised (besides well-controlled HIV) or on immunosuppressive therapy (except for steroids for COVID), advanced cancer
* Have received oral anti-rejection or immunomodulatory drugs (including TCZ) within the past 3 months
* Participating in another interleukin (IL)-6 antagonist clinical trial or other drug clinical trials (participation in COVID-19 anti-viral trials may be permitted if approved by Medical Monitor)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 10 x upper limit of normal (ULN) detected within 24 hours at screening (according to local laboratory reference ranges)
* Absolute neutrophil count (ANC) < 1000/uL at screening (according to local laboratory reference ranges)
* Platelet count < 50,000/uL at screening (according to local laboratory reference ranges)
* Pregnant or breastfeeding, or positive pregnancy test in a pre-dose examination
* Treatment with an investigational drug within 5 half lives or 30 days (whichever is longer) of randomization (investigational COVID-19 antivirals may be permitted if approved by Medical Monitor)
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Any history of Diverticulitis or GI perforation
* Use of systemic corticosteroids unless on a stable chronic dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (44):
- United States (32):
  - Banner - University Medical Center Phoenix; In-Patient Pharmacy, Phoenix, Arizona
  - Univ of AZ Coll of Med, Tucson, Arizona
  - El Centro Regional Medical Center, El Centro, California
  - eStudySite, La Mesa, California
  - Highland Hospital Oakland, Oakland, California
  - St. Joseph'S Hospital, Orange, California
  - San Leandro Hospital; Inpatient Pharmacy, San Leandro, California
  - Larkin Community Hospital Palm Springs Campus (Hialeah), Hialeah, Florida
  - Miami Veterans Administration Healthcare System - NAVREF, Miami, Florida
  - University of Miami Pulmonary, Miami, Florida
  - Larkin Community Hospital, South Miami, Florida
  - St. Lukes Boise Medical Center, Boise, Idaho
  - Ochsner Clinic, New Orleans, Louisiana
  - Holy Cross Germantown Hospital, Germantown, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - St. Joseph'S Regional Medical Center, Paterson, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - SUNY Downstate Medical Center., Brooklyn, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Flushing Hospital, Flushing, New York
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Harlem Hospital, New York, New York
  - Canton-Potsdam Hospital, Potsdam, New York
  - St. Barnabas Hospital, The Bronx, New York
  - Novant Health Presbyterian Medical Center (Presbyterian Hospital), Charlotte, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Valley Baptist Medical Center, Harlingen, Texas
  - Michael E Debakey VA Medical Center, Houston, Texas
  - McAllen Medical Center, McAllen, Texas
  - Sentara Medical Group, Virginia Beach, Virginia
- Brazil (3):
  - Hospital E Maternidade Celso Pierro PUCCAMP, Campinas, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos CEMEC FMABC, São Bernardo do Campo, São Paulo
  - BR Trials - Pesquisa Clínica, São Paulo, São Paulo
- Aga Khan University Hospital, Nairobi, Kenya
- Mexico (2):
  - Hospital General de Culiacan, Culiacán
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
- Peru (5):
  - Hospital Militar Central, Jesus Maria
  - Hospital Nacional Sergio E. Bernales, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Hospital Nacional Hipolito; Unanue, Lima
  - Hospital Maria Auxiliadora, Lima
- George Provincial Hospital, George, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Salama C, Han J, Yau L, Reiss WG, Kramer B, Neidhart JD, Criner GJ, Kaplan-Lewis E, Baden R, Pandit L, Cameron ML, Garcia-Diaz J, Chavez V, Mekebeb-Reuter M, Lima de Menezes F, Shah R, Gonzalez-Lara MF, Assman B, Freedman J, Mohan SV. Tocilizumab in Patients Hospitalized with Covid-19 Pneumonia. N Engl J Med. 2021 Jan 7;384(1):20-30. doi: 10.1056/NEJMoa2030340. Epub 2020 Dec 17. PMID 33332779
- [Derived] Tleyjeh IM. The Misleading "Pooled Effect Estimate" of Crude Data from Observational Studies at Critical Risk of Bias: The Case of Tocilizumab in Coronavirus Disease 2019 (COVID-19). Clin Infect Dis. 2021 Jun 15;72(12):e1154-e1155. doi: 10.1093/cid/ciaa1735. No abstract available. PMID 33201228

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received one IV infusion of TCZ in addition to SOC with up to one additional infusion.
- Placebo: Participants received one intravenous (IV) infusion of placebo, in addition to SOC, with up to one additional infusion.
Period: Overall Study
Arm/Group | Tocilizumab | Placebo
Started | 249 | 128
Completed | 225 | 115
Not Completed | 24 | 13
Not completed — Death | 24 | 11
Not completed — Transferred to a different facility for care | 0 | 2

BASELINE CHARACTERISTICS:
Population: mITT population = all randomized participants who received study treatment, grouped according to the treatment assigned at randomization. Participants not receiving study treatment were excluded from analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 249 | 128 | 377
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (14.3) | 55.6 (14.9) | 55.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 55 | 154
  Male | 150 | 73 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 143 | 68 | 211
  Not Hispanic or Latino | 106 | 60 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 52 | 25 | 77
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 35 | 22 | 57
  White | 134 | 65 | 199
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 19 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Proportion of Participants Who Died or Required Mechanical Ventilation by Day 28
Description: Cumulative proportion is measured as a percentage of participants meeting the endpoint.
Time Frame: Up to Day 28
Population: mITT population = all randomized participants who received study treatment, grouped according to the treatment assigned at randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Percentage of Participants | 12.04 [8.52 to 16.86] | 19.26 [13.34 to 27.36]

2. Secondary Outcome: Time to Hospital Discharge or "Ready for Discharge" (as Evidenced by Normal Body Temperature and Respiratory Rate, and Stable Oxygen Saturation on Ambient Air or >/= 2 Liters (L) Supplemental Oxygen)
Time Frame: Up to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Days | 6.0 [6.0 to 7.0] | 7.5 [7.0 to 9.0]

3. Secondary Outcome: Time to Improvement of at Least 2 Categories Relative to Baseline on a 7-Category Ordinal Scale of Clinical Status
Description: Clinical status was assessed using a 7-category ordinal scale:
  1. - Discharged (or "ready for discharge" as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient air or </=2 liters supplemental oxygen)
  2. - Non- intensive care unit (ICU) hospital ward (or "ready for hospital ward") not requiring supplemental oxygen
  3. - Non-ICU hospital ward (or "ready for hospital ward") requiring supplemental oxygen
  4. - ICU or non-ICU hospital ward, requiring non-invasive ventilation or high-flow oxygen
  5. - ICU, requiring intubation and mechanical ventilation
  6. - ICU, requiring extracorporeal membrane oxygenation (ECMO) or mechanical ventilation and additional organ support
  7. - Death
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Days | 6.0 [6.0 to 7.0] | 7.0 [6.0 to 9.0]

4. Secondary Outcome: Time to Clinical Failure, Defined as the Time to Death, Mechanical Ventilation, ICU Admission, or Withdrawal (Whichever Occurred First)
Time Frame: Up to Day 28
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Days | NA [NA to NA] — Value is NA due to an insufficient number of participants with the event. | NA [NA to NA] — Value is NA due to an insufficient number of participants with the event.

5. Secondary Outcome: Mortality Rate by Day 28
Time Frame: Up to Day 28
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Percentage of Participants | 10.4 [7.2 to 14.9] | 8.6 [4.9 to 14.7]

6. Secondary Outcome: Clinical Status on 7-Category Ordinal Scale at Day 28
Description: as for outcome 3
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 249 | 128
Percentage of participants
  1 | 85.9 | 82.8
  2 | 0.4 | 1.6
  3 | 2.0 | 0.8
  4 | 0.4 | 0.8
  5 | 0.8 | 3.9
  6 | 0 | 1.6
  7 | 10.4 | 8.6

7. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to Day 60
Population: Safety evaluable population = all participants who received any amount of study drug, grouped according to the treatment first received rather than by the treatment assigned at randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 250 | 127
Percentage of participants | 50.8 | 52.8

ADVERSE EVENTS:
Time Frame: Up to Day 60
Description: The safety evaluable population included all participants who received any amount of study drug, grouped according to the treatment first received rather than by the treatment assigned at randomization.
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 29/250 | 15/127
Serious Adverse Events (participants affected / at risk) | 38/250 | 25/127
Other Adverse Events (participants affected / at risk) | 28/250 | 8/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=250) | Placebo (N=127)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 5 (5) | 3 (3)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=250) | Placebo (N=127)
Constipation (Gastrointestinal disorders) | 16 (16) | 4 (4)
Anxiety (Psychiatric disorders) | 15 (15) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT04372186/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT04372186/SAP_001.pdf